CLINICAL TRIAL: NCT05005585
Title: Vestibular Socket Therapy With Simultaneous Implant Placement Versus Contour Augmentation With Early Implant Placement in Fresh Extraction Sockets : A Randomized Clinical Trial
Brief Title: Vestibular Socket Therapy With Simultaneous Implant Placement Versus Contour Augmentation With Early Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Iman Abd-ElWahab Radi, PhD, Professor of Prosthodontics, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: vst versus contour aug.
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Loss of Teeth Due to Extraction
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: VST with immediate implant placement versus contour augmentation with early implant placement in fresh extraction sockets in esthetic zone.
Who Masked: Outcomes Assessor
Masking Description: outcome assessor isnt involved in the intervension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vestibuler socket therapy (Experimental): immediate implant placement in esthatic zone with final crown placement after 2 months with VST technique
  Interventions: Procedure: immediate implant
- contour augmentation (Experimental): Early implant placement in esthatic zone with contour augmentation and final crown after 3 months of implant placement
  Interventions: Procedure: immediate implant

INTERVENTIONS:
Procedure: immediate implant — immediate implant placement with VST technique versus early implant placement with contour augmentation technique

SUMMARY:
immediate implant placement with VST technique versus early implant placement with contour augmentation in fresh extraction sockets in the esthetic zone.

DETAILED DESCRIPTION:
comparing VST technique with immediate implant placement that end up with final crown after 2 months with contour augmentation with early implant placement after 4- 8 weeks of soft tissue healing , then after 3 months final crown delivery both in fresh extraction sockets in the esthetic zone .

ELIGIBILITY:
Inclusion Criteria:

Non-restorable maxillary teeth in the esthetic zone

Intact adjacent teeth

Adequate palatal and apical bone that allows achieving implant primary stability.

Compromised sockets type II defect (Nicolas Elian 2007)

≥18 years

Systemically healthy patients

Exclusion Criteria:

Extraction sockets with acute or chronic infection or with adjacent infected teeth

Heavy Smokers > than 10 cigarettes daily

Cancer patients undergoing radiotherapy or chemotherapy during or within the last 6 months.

Unmotivated patients to maintain adequate oral hygiene to follow up.

Patients with physical disabilities that could affect follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 12 months
  If there is no pain or tenderness on use, no mobility, no history of exudates and radiographic bone loss is less than 2 mm from initial surgery implant the implant is considered successful

SECONDARY OUTCOMES:
Changes in the height and thickness of the labial plate of bone | 12 months
  will be measured by superimposing CBCT images obtained at the baseline (time of tooth extraction) and those after 12 months postimplant placement.
Changes in soft tissue height | 12 months
  were identified midfacially and at the apex of the mesial and distal papillae by superimposing the STL (Standard Triangle Language) files of the models, obtained via IOS, at the baseline (of the unrestorable tooth) with those after 12 months of implant insertion

CONTACTS AND LOCATIONS:
Overall Officials: Iman Radi, PHD, Study Director — Professor of prosthodontics; AbdelSalam ElAsakry, BDS, Study Director — Private Practice
Locations (3):
- Egypt (3):
  - Faculty of dentistry Cairo university, Cairo, Giza Governorate
  - Faculty of dentistry, Cairo, Manial
  - Iman AbdelWahab Radi, Cairo